CLINICAL TRIAL: NCT04327622
Title: Prevalence and Risk Evaluation of Diabetic Complications of the Foot in A Large Canadian Population
Acronym: PEDAL
Status: Completed | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: PEDAL
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Foot Deformities; Onychauxis; Neuropathy, Diabetic; Hyperkeratosis; Onychomycosis; Foot Ulcer, Diabetic
Keywords: Diabetes; Observational Study; Diabetic Foot Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Foot Deformities; Nails, Malformed; Diabetic Neuropathies; Keratoderma, Palmoplantar, Epidermolytic; Onychomycosis; Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to assess foot complications among patients with diabetes in Canada, using patient data collected during diabetes foot assessments performed by the LMC Chiropody Team between February 27, 2018 and April 17, 2019.

DETAILED DESCRIPTION:
Among patients with diabetes, one of the major causes of increased morbidity and mortality include lower-extremity complications. Patients who have peripheral neuropathy and peripheral arterial disease are at risk of developing foot ulcers and infection, which can lead to lower-extremity amputations. Adults with diabetes in Canada are 20 times more likely to be hospitalized for a nontraumatic lower limb amputation than adults without diabetes. Thus, the prevention, education and early treatment of diabetes foot complications are an important component of caring for patients living with diabetes.

In addition to neuropathy and peripheral arterial disease, risk factors for developing foot ulcers include increased levels of glycated hemoglobin, onychomycosis, microvascular complications, previous foot ulcer or amputation, structural deformity, and limited joint mobility. To the best of our knowledge, the prevalence of foot complications, such as onychomycosis, and the association of diabetes foot complications with glycemic control and other diabetes risk factors, has not been assessed before in a large sample of Canadian patients. To better understand foot complications among patients with diabetes in Canada, the investigators will retrospectively examine patient data collected during diabetes foot assessments performed by the LMC Chiropody Team. The LMC Chiropody Team is part of LMC Diabetes & Endocrinology, which is one of the largest endocrine practice groups globally.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of type 1 or type 2 diabetes
* Under the care of an endocrinologist at LMC
* Diabetes foot assessment was performed by the LMC Chiropody Team
* Informed consent to use patient medical record data for research purposes was provided

Exclusion Criteria:

* Prior diabetes foot assessment by an LMC chiropodist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes at LMC Diabetes & Endocrinology, who were provided with an initial diabetes foot assessment supported by funding from Bausch Canada. The diabetes foot assessments were performed by the LMC Chiropody Team at seven of the Ontario LMC clinics between February 27, 2018 and April 17, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 5084 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of diabetes foot complications: foot ulcer | 24-hours
  Proportion of patients diagnosed with a foot ulcer
Prevalence of diabetes foot complications: onychocryptosis | 24-hours
  Proportion of patients with onychocryptosis
Prevalence of diabetes foot complications: onychomycosis | 24-hours
  Proportion of patients with onychomycosis
Prevalence of diabetes foot complications: onychauxis | 24-hours
  Proportion of patients with onychauxis
Prevalence of diabetes foot complications: hyperkeratosis | 24-hours
  Proportion of patients with hyperkeratosis
Prevalence of diabetes foot complications: foot deformities | 24-hours
  Proportion of patients with foot deformities
Prevalence of diabetes foot complications: neuropathy risk | 24-hours
  Risk for neuropathy will be measured using the modified Toronto Clinical Neuropathy Score (mTCNS)

SECONDARY OUTCOMES:
Diabetes foot assessment risk group | 24-hours
  Diabetes foot assessment risk group will be determined according to International Diabetes Federation (IDF) recommendations. Proportion of patients with low, moderate, high and very high risk will be reported.
Association between foot risk variables and the presence of a foot ulcer | 24-hours
  Risk factors that are associated with foot ulcers in our patient cohort with diabetes will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Aronson, MD, Principal Investigator — LMC Healthcare
Locations (1):
- LMC Healthcare, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Undecided